CLINICAL TRIAL: NCT01937169
Title: Targeting Dopamine Therapy in RLS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TASMC-13-TH-0416-CTIL
Record Dates: First submitted 2013-09-03; First posted 2013-09-09 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2013-12

CONDITIONS: Restless Legs Syndrome
MeSH Terms: conditions — Restless Legs Syndrome | interventions — Levodopa

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Drug + motor task (Experimental): Each participant will undergo physical examination by an doctor. Then, the participant will receive the Fitbit device with instructions for proper use. The next stages will take place at the participant's home environment.
  Each participant will monitor motor activity in hours prior to sleep and at night for assessing baseline activity level. After 3 nights of monitoring, each participant will be administered with a quarter of a Dopicar pill (4th night) and half a Dopical pill (5th night), measuring different dose effect on motor activity during sleep.This group will be administered with a quarter of a Dopicar pill, 1 hour prior to sleep. After 15 minutes, participants in this group will perform a motor task (e.g., walking) for 30 minutes.
  Interventions: Behavioral: Motor Task; Drug: Levodopa tablet
- Placebo + motor task (Placebo Comparator): Each participant will undergo physical examination by an doctor. Then, the participant will receive the Fitbit device with instructions for proper use. The next stages will take place at the participant's home environment.
  Each participant will monitor motor activity in hours prior to sleep and at night for assessing baseline activity level. After 3 nights of monitoring, each participant will be administered with a quarter of a Dopicar pill (4th night) and half a Dopical pill (5th night), measuring different dose effect on motor activity during sleep. This group will be administered with a quarter of a Placebo pill, 1 hour prior to sleep. After 15 minutes, participants in this group will perform a motor task (e.g., walking) for 30 minutes.
  Interventions: Behavioral: Motor Task; Drug: Placebo pill
- Dopicar + Sham task (Sham Comparator): Each participant will undergo physical examination by an doctor. Then, the participant will receive the Fitbit device with instructions for proper use. The next stages will take place at the participant's home environment.
  Each participant will monitor motor activity in hours prior to sleep and at night for assessing baseline activity level. After 3 nights of monitoring, each participant will be administered with a quarter of a Dopicar pill (4th night) and half a Dopical pill (5th night), measuring different dose effect on motor activity during sleep. This group will be administered with a quarter of a Dopicar pill, 1 hour prior to sleep. After 15 minutes, participants in this group will perform a non-motor task (e.g., crossword puzzle) for 30 minutes.
  Interventions: Drug: Levodopa tablet; Behavioral: Sham non-motor task

INTERVENTIONS:
Behavioral: Motor Task — A motor task executed for 30 minutes after drug adminidtration
  Arms: Drug + motor task; Placebo + motor task
Drug: Levodopa tablet
  Arms: Dopicar + Sham task; Drug + motor task
Behavioral: Sham non-motor task — A non-motor task )sham condition) will be executed for 30 minutes after drug adminidtration
  Arms: Dopicar + Sham task
Drug: Placebo pill
  Arms: Placebo + motor task

SUMMARY:
Neurons in the brain require blood and oxygen for proper function. The term "neurovascular coupling" has been postulated in the 19th century by Roy & Sherrington referring to increased blood flow to active neurons. The rationale of this research relies on the neurovascular coupling, suggesting that increased blood flow to active regions on the brain should supply not only more blood, but also more of a pharmacological agent present in the blood system at the time. Thus, active regions should be affected by the agent (=drug) to a greater extent.

In the present study we focus on the dopaminergic system, critical in many functions such as cognition, response to stimuli and movement. One of the well-known dopaminergic pathways in the brain is the nigrostriatal pathway, mediating motor function. In this research, we intend to examine the effects of coupling functional activation in this pathway with a dopaminergic agent, Carbidopa/Levodopa, on symptoms of Restless Leg Syndrome (RLS). RLS is characterized by an irresistible urge to move the limbs (i.e. Akathisia), and results most prominently by a significant decrease in the quality of sleep. Our research focuses on this symptom of RLS to examine the effect of coupling brain activation and drug treatment.

The first line of treatment in RLS is dopaminergic drugs. These drugs increase dopamine levels in motor pathways, and our research will aim to couple activation in the nigrostriatal motor pathway with dopaminergic treatment in RLS. Functional activation will be achieved with a simple motor task, known to elicit activation in the nigrostriatal pathway. We hypothesize that the drug will act upon the pre-activated motor system, and that this coupling between brain activation and drug treatment will ameliorate sleep-related symptoms of RLS, compared with treating these symptoms solely with a dopaminergic drug and compared with using a non-motor task.

ELIGIBILITY:
Inclusion Criteria:

RLS diagnosis according the common clinical criteria No known neurological illnesses No known Kidney illnesses No known iron deficiency No history of drug or alcohol use

Exclusion Criteria:

Regular drug treatment Use of a psychotropic substance in the two weeks prior to the study Auditory or Visual impairment Psychiatric history Neurological illness Chronic Kidney illness Obstructive Sleep Apnea (OSA) Dopaminergic drug intolerance or sensitivity Glaucoma Melanoma or Pre-Melanoma (current or previous) Pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-01; Primary Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Efficacy | 1 week
  Nighttime measures of motor activity will be used to assess the efficacy of treatment intervention

SECONDARY OUTCOMES:
reported efficacy | 1 week
  Participant's reports of the quality of sleep will be recorded

CONTACTS AND LOCATIONS:
Locations (1):
- Tel Aviv Sourasky Medical Center, Tel Aviv, N/A = Not Applicable, Israel